CLINICAL TRIAL: NCT06192251
Title: Complete Lifestyle Medicine Intervention Program (CLIP)
Brief Title: Complete Lifestyle Medicine Intervention Program
Acronym: CLIP
Status: Recruiting | Type: Observational
Sponsor: Northern Ontario School of Medicine (Other)
Responsible Party: Principal Investigator, Lisa Allen, Research Coordinator, Director of Reserach, Parry Sound, Huntsville and Bracebridge, Northern Ontario School of Medicine
Other Study IDs: CLIP
Record Dates: First submitted 2023-12-15; First posted 2024-01-05 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: High Cholesterol; Diabetes; Obesity; Hypertension; Heart Diseases
MeSH Terms: conditions — Hypercholesterolemia; Diabetes Mellitus; Obesity; Hypertension; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Weekly classes of pillars of lifestyle medicine, monthly sessions with dietician, Lifestyle Medicine physician,kinesiologist and health coach
  Interventions: Behavioral: Lifestyle Medicine

INTERVENTIONS:
Behavioral: Lifestyle Medicine — Education and support for lifestyle modification to improve health conditions

SUMMARY:
This project will use a mixed design and will be conducted at the West Parry Sound Health Centre. Based on similar studies there is an expected 10% drop-out rate so 20 participants per group will be invited to aim to have 15 finish. Total participants invited over the two-year study will be 40. The participants will be followed over a Complete 6-month Lifestyle medicine Intervention Program (CLIP) involving a collaboration between physicians, health coach, registered dietitians, and kinesiology. The CLIP will cover the 6 pillars of lifestyle medicine in 12-14 fundamentals of lifestyle medicine group classes.

DETAILED DESCRIPTION:
Participants will have the option of a hybrid platform to ensure equal access. Participants will attend (virtually or in person) a weekly lecture on Lifestyle Medicine Pillars for 16 weeks followed by a weekly exercise program for 8 weeks. This program was inspired by the research team of Albert et al 2022.

The eligibility criteria for participation in the lifestyle medicine program include adults with chronic diseases such as

* prediabetes,
* type 2 diabetes,
* pre-hypertension,
* systemic hypertension,
* heart disease, dyslipidemia,
* and/or excess weight (BMI ≥ 25 (42)).

Patients will be invited through referral by their physicians, email by local heart disease and diabetes foundation, mail-out by nurse practitioner and community health teams. Metrics:

Participants will be evaluated using validated pre-and post intervention validated surveys provided by the American College of Lifestyle Medicine, The Lifestyle Assessment Short Form. Added to the validated survey included questions on demographic characteristics including gender, age, race and ethnicity, language use, education, health insurance marital status. Participants will complete The Well-being Assessment and Lifestyle Medicine Survey (American College of Lifestyle Medicine)

ELIGIBILITY:
Inclusion Criteria:

* prediabetes,
* type 2 diabetes,
* pre-hypertension,
* systemic hypertension,
* heart disease, dyslipidemia,
* and/or excess weight (BMI ≥ 25 (42)).

Exclusion Criteria:

* Healthy participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligibility criteria for participation in the lifestyle medicine program include adults with chronic diseases such as prediabetes, type 2 diabetes, pre-hypertension, systemic hypertension, heart disease, dyslipidemia, and/or excess weight (BMI ≥ 25 (42)). Patients will be invited through referral by their physicians, email by local heart disease and diabetes foundation, mail-out by nurse practitioner and community health teams
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-08-06 (Estimated); Study Completion 2026-11-06 (Estimated)

PRIMARY OUTCOMES:
Participant Feedback | 1 month
  Collect pre-and post intervention survey responses using the validated Lifestyle Medicine Scales (The Lifestyle Assessment Short Form) and The Well-being Assessment and Lifestyle Medicine Survey)
Participant Feedback | 1 month
  Collect pre-and post intervention survey responses using the validated Lifestyle Medicine Scales (The Well-being Assessment Survey)
Participant Feedback | 1 month
  Collect pre-and post intervention survey responses using the validated Lifestyle Medicine Scales (Lifestyle Medicine Survey)

SECONDARY OUTCOMES:
Participant Feedback | 6 months
  Participants will be invited to participate in focus groups at the end of the 22 week intervention to share their opinions about the material covered, how the study could be improved and general feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Rheaume, MD, Study Chair — Laval
Locations (1):
- West Parry Sound Health Centre, Parry Sound, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data will be shared

REFERENCES:
- [Derived] Patel K, Allen L, Boucher K, Fedele M, Fong D, Kumar S, Lavigne D, Marin-Couture E, Partyka-Sitnik M, Rietze N, Smith-Turchyn J, Juneau M, Rheaume C. Complete Lifestyle Medicine Intervention Program-Ontario: Implementation Protocol for a Rural Study. JMIR Res Protoc. 2024 Dec 31;13:e59179. doi: 10.2196/59179. PMID 39740215